CLINICAL TRIAL: NCT06224231
Title: Patient Survey 2024 and Following Years as a Tool to Quality Assurance and Quality Improvement - CharitéCentrum for Anesthesiology and Intensive Care Medicine 007, Charité - Universitätsmedizin Berlin
Brief Title: Patient Survey as a Tool to Quality Assurance and Quality Improvement 2024
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the CharitéCentrum for Anesthesiology and Intensive Care Medicine 007, Charite University, Berlin, Germany
Other Study IDs: QM-Patient survey 2024
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One goal of the investigators of the Department of Anesthesiology and Intensive Care Medicine CCM/CVK, Charité - Universitätsmedizin Berlin is a continuous improvement in the quality of care to the patients. One focus is the freezing preoperatively during surgery, and on the follow-up study to assess the perceived waiting times in the anesthesiology outpatient clinic.

The project aims to quality assurance and quality improvement of the CharitéCentrum for Anesthesiology and Intensive Care Medicine 007, Charité - Universitätsmedizin Berlin .

DETAILED DESCRIPTION:
The primary objective of the survey is to assess the entire perioperative care with particular focus on the development of perceived waiting times in the anesthesiology outpatient clinic, re-evaluation of the preoperative freezing the preoperative thirst, pain, nausea and vomiting after surgery (PONV prophylaxis).

The survey will be repeated in a three-year interval (approximately 1000 - 2000 patients per survey) to monitor and improve the quality of the CharitéCentrum for Anesthesiology and Intensive Care Medicine 007, Charité - Universitätsmedizin Berlin from the patient point of view.

In order to achieve a meaningful data collection, a response rate of 50 percent should be achieved.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients who underwent a procedure in anesthesia and willing to take part in the Survey
* aged >= 1 years

Exclusion Criteria:

* unconscious patients,
* refusal by patient / parents

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients who underwent a procedure in anesthesia
Sampling Method: Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | Time during hospital stay, an average of 2 weeks
  Patient satisfaction with the care provided by the staff of the CC07; Measurement of satisfaction: Yes/No/Partly

SECONDARY OUTCOMES:
Campus | Time in the outpatient clinic of anesthesia, an average of 1 hour
  Campus: CCM or CVK or CBF
Waiting time in the premedication visit | Time in the outpatient clinic of anesthesia, an average of 1 hour
  Measurement of waiting time: < 15 minutes, 15-30 minutes, 30-60 minutes, > 60 minutes
Friendliness of the staff during the premedication visit | Time in the outpatient clinic of anesthesia, an average of 1 hour
  Measurement of friendliness: Yes/No/Partly
Information provided during the premedication visit by the anesthetist | Time in the outpatient clinic of anesthesia, an average of 1 hour
  Measurement of Information: Yes/No/Partly
Response to questions during the premedication visit | Time in the outpatient clinic of anesthesia, an average of 1 hour
  Response to questions is measured: Yes/No/Partly
Fear reduction during the premedication visit | Time in the outpatient clinic of anesthesia, an average of 1 hour
  Fear reduction is measured: Yes/No/Partly
Information provided during the premedication visit by educational films | Time in the outpatient clinic of anesthesia, an average of 1 hour
  Measurement of information by educational films: Yes/No/Partly/No film
Compliance with the planned start of the operation | Time in the operation room before start of anesthesia, an average of 30 minutes
  Measurement of compliance with the start of the operation: Yes/No
Friendliness of staff | Time in the operation room before start of anesthesia, an average of 30 minutes
  Measurement of friendliness: Yes/No/Partly
Fear | Time in the operation room before start of anesthesia, an average of 30 minutes
  Fear measured: Yes, very much/Yes, but not much/No fear /Partly
Thirst | Time in the operation room before start of anesthesia, an average of 30 minutes
  Thirst measured: Yes, very much/Yes, but not much/No thirst/Partly
Pain | Time in the operation room before start of anesthesia, an average of 30 minutes
  Pain measured: Yes, strong pain/Yes, but not strong/No pain/Can't remember
Sufficient pain treatment | Time in the operation room before start of anesthesia, an average of 30 minutes
  Sufficient pain treatment measured: Yes, sufficiently treated/ Treated, but not sufficiently/Not treated/No pain/No treatment wanted/Partly
Shivering | Time in the operation room before start of anesthesia, an average of 30 minutes
  Shivering is measured: Yes, strong/Yes, but not strong/No shivering/Partly
Sufficient therapy in case of shivering | Time in the operation room before start of anesthesia, an average of 30 minutes
  Sufficient therapy in case of shivering is measured: Yes, sufficiently treated/ Treated, but not sufficiently/Not treated/No shivering/No treatment wanted/ Partly
Friendliness of staff | Time in the intensive care unit or post anesthesia care unit, an average of 3 days
  Friendliness is measured: Yes/No/Partly
Post-operative nausea and vomiting (PONV) | Time in the intensive care unit or post anesthesia care unit, an average of 3 days
  Measurement of PONV: nausea/vomiting/nausea and vomiting/neither nor
Sufficient therapy in case of PONV | Time in the intensive care unit or post anesthesia care unit, an average of 3 days
  Sufficient therapy is measured: Yes, sufficiently treated/ Treated, but not sufficiently/Not treated/No PONV/No treatment wanted/Partly
Pain intensity | Time in the intensive care unit or post anesthesia care unit, an average of 3 days
  Pain intensity is measured by likert scale: strong, moderate, low, none
Sufficient therapy in case of pain | Time in the intensive care unit or post anesthesia care unit, an average of 3 days
  Sufficient therapy is measured: Yes, sufficiently treated/ Treated, but not sufficiently/Not treated/No pain/No treatment wanted/Partly
Shivering | Time in the intensive care unit or post anesthesia care unit, an average of 3 days
  Sufficient therapy in case of shivering is measured: Yes/No/Partly
Sufficient therapy in case of shivering | Time in the intensive care unit or post anesthesia care unit, an average of 3 days
  Sufficient therapy in case of shivering is measured: Yes, sufficiently treated/ Treated, but not sufficiently/Not treated/No shivering/No treatment wanted/Partly
Post-operative nausea and vomiting (PONV) | Time during hospital stay, an average of 2 weeks
  Measurement of PONV: nausea/vomiting/nausea and vomiting/neither nor
Regional anaesthesia | Time during hospital stay, an average of 2 weeks
  Measured: Yes / No
Satisfaction with regional anaesthesia | Time during hospital stay, an average of 2 weeks
  Measurement of satisfaction: Yes/No/Partly
In case of need choosing of regional anaesthesia again | Time during hospital stay, an average of 2 weeks
  Measurement of choosing again: Yes/No/Perhaps
Satisfaction of care through pain service | Time during hospital stay, an average of 2 weeks
  Measurement of care through pain service: Yes/No/Partly
Recommendation of medical care (provided by the staff from CC07) | Time during hospital stay, an average of 2 weeks
  Measurement of recommendation: Yes/No/Partly
Atmosphere | Time in the intensive care unit or post anesthesia care unit, an average of 3 days
  Measurement of atmosphere: calm/busy/can´t remember
Postoperative fear | Time in the intensive care unit or post anesthesia care unit, an average of 3 days
  Measurement of fear: Yes, very much/Yes, but not much/No fear
Postoperative pain | Time during hospital stay, an average of 2 weeks
  Pain intensity is measured by likert scale: strong, moderate, low, none
Sufficient therapy in case of pain | Time during hospital stay, an average of 2 weeks
  Sufficient therapy is measured: Yes, sufficiently treated/ Treated, but not sufficiently/Not treated/No pain/No treatment wanted/Partly
Postoperative patient controlled analgesia | Time during hospital stay, an average of 2 weeks
  Measurement: Yes/No/I don´t know
Choosing of Patient controlled anesthesia | Time during hospital stay, an average of 2 weeks
  Question: Would you choose patient controlled anesthesia again? Answer: Yes/No/Maybe

OTHER OUTCOMES:
Postoperative stay | Time during hospital stay, an average of 2 weeks
  Postoperative stay is measured by: in post anesthesia care unit/intensive care unit/unknown

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte and Campus Virchow-Klinikum, Charité - Universitaetsmedizin Berlin, Berlin, State of Berlin
  - Department of Anesthesiology and Intensive Care Medicine (CBF), Charité - Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No